CLINICAL TRIAL: NCT01505218
Title: Patient-controlled Propofol Sedation for Endoscopic Retrograde Cholangiopancreatography
Brief Title: Propofol Patient-controlled Sedation for Endoscopic Retrograde Cholangiopancreatography
Acronym: PER-projekt
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Linkoeping (Other)
Responsible Party: Principal Investigator, Lena Nilsson, MD, PhP, senior consultant, University Hospital, Linkoeping
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PER 2010/232-31
Record Dates: First submitted 2011-12-13; First posted 2012-01-06 (Estimated); Last update posted 2020-11-09 (Actual); Status verified 2015-12

CONDITIONS: Endoscopic Retrograde Cholangiopancreatography
Keywords: Sedation; propofol; patient-controlled; safety

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Propofol sedation by nurse anaesthetist (Active Comparator): Nurse anaesthetists managed infusion of propofol 10 mg/ml at doses of 0.2 - 0.8 ml/kg during ERCP. The target of moderate sedation was achieved within 5 minutes from start of the sedation.
  Interventions: Drug: Propofol sedation by nurse anaesthestist
- Patient-controlled propofol sedation (Active Comparator): Self-administration of propofol via patient-controlled sedation pump (CME...). No programmed lock-out period, no dose limit or background infusion. 5 mg propofol/effectuated demand from the patients. Capacity of the pump was 6 possible doses per minute.
  Before start of ERCP the patients were allowed to sedate themselves to a sense of heavy tiredness.
  Interventions: Drug: Patient-controlled propofol sedation
- Midazolam sedation by the ERCP-team (No Intervention): Midazolam doses for sedation during ERCP. Initial dose of 2-3 mg and after ERCP start, 1-2 mg as additional doses. Maximum total dose 6-8 mg. ERCP performing doctor is responsible for dose ordination.

INTERVENTIONS:
Drug: Propofol sedation by nurse anaesthestist — Propofol (10 mg/ml) is a short-acting, intravenously administered hypnotic agent used for light-moderate-deep sedation.
  Patient-controlled sedation: self-administration of propofol boluses of 5 mg with zero lock-out time. Administration time for the pump was 12 sec, equivalent to maximum delivery of 25 mg of propofol per minute.
  Propofol sedation by nurse anaesthetists:
  Arms: Propofol sedation by nurse anaesthetist
Drug: Patient-controlled propofol sedation — Propofol (10 mg/ml) is a short-acting, intravenously administered hypnotic agent used for light-moderate-deep sedation.
  Self-administration of propofol via patient-controlled sedation pump (CME T-34L PCA). No programmed lock-out period, no dose limit or background infusion. 5 mg propofol/effectuated demand from the patients. Capacity of the pump was 6 possible doses per minute.
  Before start of ERCP the patients were allowed to sedate themselves to a sense of heavy tiredness.
  Arms: Patient-controlled propofol sedation

SUMMARY:
Propofol sedation with opioids is used for endoscopic retrograde cholangiopancreatography (ERCP). Combination of sedatives and opioids is associated with increased morbidity/mortality. Delivery of only propofol using a patient-controlled delivery system (patient-controlled sedation, PCS) could be an alternative for this purpose. Comparative studies with PCS for ERCP are few. Therefore, the main objective of this randomized controlled trial was to compare propofol PCS to sedation managed by nurse anaesthetists during ERCP.

ELIGIBILITY:
Inclusion Criteria:

* Need for ERCP
* Able to speak and read swedish

Exclusion Criteria:

* Allergy to propofol
* Severe cardiopulmonary disease (ASA IV)
* Confusion or dementia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 281 (Actual)
Dates: Start 2010-10; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
treatability | one day (per-procedural)
  Registration of number of failures (where procedure is interrupted as a result of inadequate sedation). Comparison data between propofol PCS and nurse anaesthetists sedation using propofol and control group (midazolam).

SECONDARY OUTCOMES:
Vital signs | one and a half year
  Vital signs and interventions of nurse anaesthetists. Data on heart rate, blood pressure, peripheral oxygen saturatuion, respiratory rate, delivery of oxygen, airway obstruction assessment, airway manipulation.

CONTACTS AND LOCATIONS:
Overall Officials: Folke Sjöberg, Professor, Study Chair — Dept of Anaesthesia and Intensive Care, Linköping University Hospital, 581 85 Linköping, Sweden
Locations (1):
- Linköping University Hospital, Linköping, Sweden